CLINICAL TRIAL: NCT04419259
Title: An Open Label Study to Evaluate the Efficacy and Tolerability of Erenumab in the Management of Persistent Redness and Flushing in Rosacea
Brief Title: Efficacy and Tolerability of Erenumab in the Management of Persistent Redness and Flushing in Rosacea
Acronym: STOP Ros
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Messoud Ashina (Other)
Collaborators: Danish Headache Center (Other); Novartis Pharmaceuticals (Industry); Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor-Investigator, Messoud Ashina, Professor, MD, PhD, DMSc, Danish Headache Center
Organization: Danish Headache Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROS031019
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Erenumab (Experimental): 30 subjects with rosacea will be allocated to receive monthly subcutaneous injections of 140 mg erenumab at three time points (week 0, week 4, week 8)
  Interventions: Drug: AMG 334

INTERVENTIONS:
Drug: AMG 334 — 30 subjects with rosacea will be allocated to receive monthly subcutaneous injections of 140 mg erenumab at three time points (week 0, week 4, week 8)
  Other Names: Erenumab

SUMMARY:
An exploratory open-label study of rosacea patients to study the efficacy and tolerability of erenumab in the prophylactic treatment of persistent redness and flushing attributed to rosacea. Approximately 30 subjects will be included in the study and receive erenumab 140 mg for three months. The study will begin June 2020 and is expected to last nine months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between ages 18 - 65 years who have suffered from rosacea for at least 12 months.
* If patient has concurrent migraine, a daily headache diary must be filled out

Criteria to be met prior to enrollment in the 4-week run-in period:

•Erythematotelangiectatic rosacea with a minimum of 15 days of either:

* PSA > 2, and/or
* Moderate, severe or extreme flushing measured by the Flushing Assessment Tool (FAST)

Exclusion Criteria:

* Systemic treatment for rosacea ended less than five half-lives or 28 days ago, whichever is longest
* Topical treatment for rosacea ended less than five half-lives or 28 days ago, whichever is longest
* Cardiovascular disease of any kind, including cerebrovascular disease
* Hypertension on the experimental day (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Hypotension on the experimental day (systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 50 mmHg)
* Ongoing psychiatric disease of any kind - unless it has been effectively treated with a stable treatment for at least 2 months.
* Anamnestic or clinical symptoms of any kind that are deemed relevant for study participation by the physician who examines the patient
* Pregnant or breastfeeding women, or women expecting to conceive during the study
* Women of childbearing potential who are unwilling to use an acceptable method of effective contraception during treatment through 16 weeks after the last dose of erenumab. Acceptable methods of effective birth control include not having intercourse (true abstinence, when this is in line with the preferred and usual lifestyle of the subject), hormonal birth control methods (pills, shots/injections, implants, or patches), intrauterine devices, surgical contraceptive methods (vasectomy with medical assessment of the surgical success of this procedure or bilateral tubal ligation), or two barrier methods (each partner must use one barrier method) with spermicide - males must use a condom with spermicide; females must choose either a diaphragm with spermicide, OR cervical cap with spermicide, OR contraceptive sponge with spermicide. Female subjects not of childbearing potential are defined as any female who: is post-menopausal by history, defined as:

  * Age ≥ 55 years with cessation of menses for 12 or more months, OR
  * Age < 55 years but no spontaneous menses for at least 2 years, OR
  * Age < 55 years and spontaneous menses within the past 1 year, but currently amenorrhoeic (e.g. spontaneous or secondary to hysterectomy), AND with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved OR Underwent bilateral oophorectomy OR Underwent hysterectomy OR Underwent bilateral salpingectomy
* Known sensitivity to any component of erenumab
* Previously randomized into an erenumab study
* Member of investigational site staff or relative of the investigator
* Unlikely to be able to complete all protocol required study visits or procedures, and/or to comply with all required study procedures to the best of the subject's and investigator's knowledge

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Effect of erenumab on days of flushing | 12 weeks
  Mean change in number of days with moderate, severe or extreme flushing from Baseline to week 12. Evaluated by the Flushing Assessment (FAST) Tool part II (moderate, severe or very severe flushing is defined as a score of 4-10 on FAST)

SECONDARY OUTCOMES:
Effect of erenumab on erythema | 12 weeks
  Mean change in erythema from Baseline to week 4, 8 and 12. Will be evaluated by Clinicians Erythema Assessment (CEA)
Effect of erenumab on quality of life: Dermatology Life Quality Index (DLQI) | 12 weeks
  Mean change in quality of life from Baseline to week 4, 8 and 12. Will be evaluated by Dermatology Life Quality Index (DLQI)
Proportion of patients that reach a 50% reduction in number of days with flushing | 12 weeks
  To evaluate the proportion of patients with at least 50% reduction in number of days with moderate, severe or extreme flushing. Evaluated by the Flushing Assessment (FAST) Tool part II (moderate, severe or very severe flushing is defined as a score of 4-10 on FAST)
Effect of erenumab on days of flushing | 8 weeks
  Mean change in number of days with moderate, severe or extreme flushing from Baseline to week 4 and 8. Evaluated by the Flushing Assessment (FAST) Tool part II (moderate, severe or very severe flushing is defined as a score of 4-10 on FAST)
Effect of erenumab on depression | 12 weeks
  Mean change in depressive symptoms from Baseline to week 4, 8 and 12. Evaluated by Hospital Anxiety and Depression Scale (HADS).
Effect of erenumab on overall rosacea symptoms | 12 weeks
  Proportion of patients with Investigator's Global Assessment (IGA) '0' or '1' with an at least 2-point reduction from baseline to week 4, 8 and 12.
Effect of erenumab on inflammatory lesions | 12 weeks
  Mean change in Inflammatory Lesion Count (ILC) from baseline to week 4, 8 and 12
Proportion of patients that reach a 50% reduction in self-assessed rosacea symptoms | 12 weeks
  Proportion of patients with at least 50% reduction in number of days with Patient's Self-Assessment (PSA) above 2 from Baseline to week 4, 8 and 12.
Effect of erenumab on self-assessed rosacea symptoms | 12 weeks
  Mean change in Patient's Self-Assessment (PSA) above 2 from Baseline to week 4, 8 and 12.
Effect of erenumab on depressive symptoms | 12 weeks
  Mean change in Quicky Inventory Depressive Symptomatology (QIDS) from Baseline to week 4, 8 and 12
Effect of erenumab on overall rosacea severity | 12 weeks
  Mean change in overall rosacea severity from Baseline to week 4, 8 and 12. Evaluated by Rosacea Area and Severity Index (RASI)
Effect of erenumab on rosacea symptoms | 12 weeks
  Mean change in rosacea symptoms from Baseline to week 4, 8 and 12. Evaluated by Rosacea Clinical Scorecard (RCS)
Effect of erenumab on rosacea-specific quality of life: Rosacea-specific Quality-of-Life index (RosaQoL) | 12 weeks
  Mean change in rosacea-specific quality of life from Baseline to week 4, 8 and 12. Evaluated by the Rosacea-specific Quality-of-Life index (RosaQoL)

OTHER OUTCOMES:
Tolerability of erenumab in patients with rosacea | 12 weeks
  To evaluate the tolerability of erenumab in patient with rosacea through assessment of adverse events at every visit from Baseline to week 4, 8 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Professor, Principal Investigator — Danish Headache Center; Nita KF Wienholtz, MD, Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wienholtz NKF, Christensen CE, Do TP, Frifelt LEW, Snellman J, Lopez-Lopez CL, Egeberg A, Thyssen JP, Ashina M. Erenumab for Treatment of Persistent Erythema and Flushing in Rosacea: A Nonrandomized Controlled Trial. JAMA Dermatol. 2024 Jun 1;160(6):612-619. doi: 10.1001/jamadermatol.2024.0408. PMID 38630457